CLINICAL TRIAL: NCT04405804
Title: A Monocentric, Open Label, Single Arm, Pilot Study on the Early Administration of Ivabradine in Children Aged >6 Months and <18 Years With Dilated Cardiomyopathy and Acute Heart Failure
Brief Title: Early Administration of Ivabradine in Children With Heart Failure
Acronym: EASI-Child
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Principal Investigator, Rachele Adorisio, MD, Bambino Gesù Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1986 / 2019; 2019-003902-29 (EudraCT Number)
Record Dates: First submitted 2020-05-26; First posted 2020-05-28 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Acute Heart Failure; Dilated Cardiomyopathy
Keywords: Ivabradine; Heart Failure; Pediatric; Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure; Cardiomyopathies | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: Simon's two-stage design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ivabradine (Experimental): Eligible patients will be given treatment with ivabradine during a titration period which will last from a minimum of 3 days to a maximum of 15 days. This will be followed by a maintenance period of another 14 days. At the end of maintenance period, primary endpoint will be assessed. After maintenance period, the patient will continue ivabradine at the same dosage during a follow-up period that will last 4 months.
  Interventions: Drug: Ivabradine 5Mg Tab

INTERVENTIONS:
Drug: Ivabradine 5Mg Tab — Initial dose of ivabradine will be:
  0.02 mg/kg/dose twice daily in patients between 6-12 months 0.05 mg/kg/dose twice daily in patients between 1-3 years and 3-18 years with a weight < 40 kg 2.5 mg/day in patients between 3-18 years with weight > 40 kg During titration phase, the dose may be increased, maintained, reduced or discontinued in accordance with titration rules. The titration rules will be adjusted on the basis of age subset and of each patient's evaluation during the titration phase, whether or not the target heart rate is reached (HR ≥ 20% compared to baseline HR) and whether or not are present bradycardia (HR should be greater than predefined by a HR threshold per age subset) and/or bradycardia-related symptoms.
  Maximum dose to be reached will be:
  0.2 mg/kg/dose twice daily in patients between 6-12 months 0.3 mg/kg/dose twice daily in patients between 1-3 years and 3-18 years with a weight < 40 kg 15 mg/day in patients between 3-18 years, weight > 40 kg

SUMMARY:
This is a monocentric, prospective, single arm, not for profit study. It is designed to study the early use of ivabradine in patients with dilated cardiomyopathy and Ejection Fraction (EF) < 45%.

DETAILED DESCRIPTION:
The study is divided into a screening and enrollment visit (V1) where eligibility for treatment will be confirmed. Ivabradine will be administered to eligible patients with increasing dosage during the titration period (TP) which will last from a minimum of 3 days to a maximum of 15 days. This will be followed by a maintenance period (MP) of the drug for a further 14 days. The follow-up period (FU) will last 4 months.

The dose of ACE inhibitors will be introduced after 72 hours of clinical stability after the introduction of titrated ivabradine at maximum dose according to protocol. The anti-aldosterone will be introduced 24 hours after the introduction of ivabradine. The diuretic will not be modified during the titration phase of the drug, unless there is clinical necessity.

During the FU ivabradine will be continued at stable dosage, in order to maintain the target heart rate (HR) reached during the maintenance phase (HR > 80 bpm, in the group of patients older than 6-12 months, or HR > 70 bpm in patients aged 1-3 years or HR > 50 bpm between 3-18 years). In all patients, the drug dose will be decreased or discontinued in case of bradycardia (HR< 80 bpm in patients 6-12 months, HR< 70 bpm in patients 1-3 years of age or HR< 60 bpm in patients 3-18 years of age) and/or symptoms related to bradycardia or for other safety reasons.

ELIGIBILITY:
Inclusion Criteria:

* Dilated cardiomyopathy defined according to the indications of the Cardiomyopathy Task Force (dilation > 2 Standard Deviations (SD) and hypokinesia);
* Class NYHA/Ross ≥ II;
* Ejection fraction < 40%;
* Patients with acute heart failure episodes (both new episode and relapse) in the last three months;
* Systolic blood pressure > 50° age and height;
* Heart rate: 6-12 months: ≥105 bpm, >1 year <3 years: ≥95 bpm, 3-5 years: ≥75 bpm, 5-18 years: >70 bpm.

Exclusion Criteria:

* Cardiogenic shock in the three months;
* Hypertrophic, restrictive or mixed cardiomyopathy;
* Acute lymphocytic myocarditis diagnosed with endomyocardial biopsy;
* Significant Valvular Pathology;
* Sinus block and congenital long QT syndrome;
* Atrial Fibrillation;
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels > 2.5 times normal, bilirubin > 3 and creatinine > 2.5 mg/dL;
* Pregnancy and/or positive pregnancy test patients;
* Hypersensitivity to the active substance or any of the excipients;
* Participation in a clinical trial in which an experimental drug was administered within 30 days or 5 half-lives of the investigational drug;
* Chronic lung disease or other clinical condition that the investigating physician believes is incompatible with the study;
* eGFR <15 mL/min/1.73 m2.

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Heart rate in b.p.m. (mean (±SD) difference from baseline) at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the response to ivabradine on heart rate after 14 days of stable therapy

SECONDARY OUTCOMES:
Heart rate in b.p.m. (mean (±SD) difference from baseline) at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the response to ivabradine on heart rate after 16 weeks of follow-up
Serum NT-proBNP in pg/mL (mean (±SD) difference from baseline) at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the response to ivabradine on serum NT-proBNP levels after 14 days of stable therapy
Serum NT-proBNP in pg/mL (mean (±SD) difference from baseline) at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the response to ivabradine on serum NT-proBNP levels after 16 weeks of follow-up
Correlation between heart rate and NT-proBNP value (Pearson correlation) at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the correlation between heart rate and serum NT-proBNP levels after 14 days of stable therapy
Correlation between heart rate and NT-proBNP value (Pearson correlation) at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the correlation between heart rate and serum NT-proBNP levels after 16 weeks of follow-up
Left ventricular function, calculated by 2D echocardiographic technique (calculation of left ventricular volume and ejection fraction - mean (±SD) difference from baseline) at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess EF, Left Ventricular End Diastolic Volume (LVEDV), Left Ventricular End Systolic Volume (LVESV) after 14 days of stable therapy
Left ventricular function, calculated by 2D echocardiographic technique (calculation of left ventricular volume and ejection fraction - mean (±SD) difference from baseline) at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess EF, LVSV, LVDV after 16 weeks of follow-up
Systolic blood pressure in mmHg (mean (±SD) difference from baseline) at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the response to ivabradine on systolic blood pressure after 14 days of stable therapy
Systolic blood pressure in mmHg (mean (±SD) difference from baseline) at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the response to ivabradine on systolic blood pressure after 16 weeks of follow-up
Use of inotropic drugs (number and % of patients who had to use inotropes at the end of maintenance) | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the need to resort to inotropic drugs within 14 days of stable ivabradine therapy
Use of inotropic drugs (number and % of patients who had to use inotropes at the end of follow-up) | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the need to resort to inotropic drugs within 16 weeks of follow-up
Number and % of dropouts at the end of maintenance | At the end of the two weeks maintenance period (17-29 days from enrollment)
  To assess the frequency of patients who exit from the study within 14 days of stable ivabradine therapy
Number and % of dropouts at the end of follow-up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the frequency of patients who exit from the study within 16 weeks of follow-up
Time (days) from start of ivabradine therapy and new episode of acute heart failure, and/or implantation of mechanical assist device at the end of follow up | At the end of the 16 weeks follow-up period (129-141 days from enrollment)
  To assess the period within main cardiological events would occur after the start of ivabradine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rachele Adorisio, MD, Principal Investigator — Bambino Gesù Hospital and Research Institute
Locations (1):
- Bambino Gesù Hospital and Research Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: No